CLINICAL TRIAL: NCT06981364
Title: Minimum Time Effect of Fish Oil on Arterial Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salisbury University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9
Record Dates: First submitted 2023-04-10; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2023-04

CONDITIONS: Arterial Stiffness
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fish Oil (Experimental): Participants randomized to fish oil will receive 4 grams of fish oil supplementation each day for the entire 6-week duration.
  Interventions: Dietary Supplement: Fish Oil
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Fish Oil

INTERVENTIONS:
Dietary Supplement: Fish Oil — Upon completion of baseline testing both groups will be instructed not to alter their normal diet and activity levels throughout the study period. Zach Townsend, an individual who will not be directly involved with the data analysis, will create a spread sheet containing the weight of the subjects and separate identifier generated via algorithm. The spread sheet will be provided to the principle and co-investigators who will partition the supplements out into 42 separate sealable bags per subject. The bags will be dispersed by Mr. Townsend to maintain the double-blind standard. Subjects will either consume 4 g/day GNC Triple Strength Fish Oil Mini, General Nutrition Corporation, Pittsburgh, PA, or placebo (dextrin) of equal volume for six weeks. They will be instructed to consume fish oil or the placebo with a glass of water at the same time every day. These protocols are similar to ones used in previous investigations1-7.

SUMMARY:
This study will seek to determine the minimum time of 4 g/day fish oil supplementation to cause a clinically significant effect on arterial stiffness. Accordingly, 30 moderately active, otherwise healthy adult subjects who are not currently taking any dietary supplementations will be recruited for the study. They will be randomized in a double-blind fashion into one of two groups: placebo group or fish oil dietary supplementation group. Subjects will either receive 4 g/day fish oil or placebo for 6 weeks. Each subject will undergo a series of baseline and follow-up tests including anthropometry, ultrasonography of the carotid artery, applanation tonometry, and blood pressure acquisition at week 0, 2, 4, and 6. Subjects will be required to maintain an activity and food log. Subjects will be asked to maintain their normal activity pattern during the study period. Repeated measures analysis of variance will be used to examine the effects of treatment and the treatment-order interaction on arterial stiffness (and other dependent variables).

DETAILED DESCRIPTION:
To determine the minimum amount of time for a clinically significant effect of daily fish oil supplementation on arterial stiffness (Figure 1). 30 subjects will be randomized in a double-blind fashion into one of two groups: placebo group or fish oil dietary supplementation group. An individual not associated with the project will monitor the randomization and blinding process. He/she will not be involved in the follow-up data collection. All analyses will be conducted in a blinded fashion.

Pre-enrollment Screening. Several study information sessions will be offered to potential subjects prior to the start of the study. These information sessions will be conducted by the principle investigator. The principle investigator will also arrange office meetings for those who have a time conflict with the information sessions. After obtaining written informed consent the potential candidates will be screened to determine if they satisfy the basic criteria of the study (see below). Candidates will be instructed to fill out a Health History Questionnaire in a place of their choosing. Candidates who successfully complete the screening process will be invited to undergo baseline and follow-up testing (see details below).

Baseline and Follow-up Testing: For baseline and follow-up testing subjects will arrive at Salisbury University Simulation Center between 8:00 and 11:00 am after a 12 hour overnight fast and having performed no vigorous physical activity for the previous 48 hours. Subjects will also be required to abstain from caffeine-containing food or beverages for the previous 24 hours. Each visit will be separated by a period of two weeks.

Visit 1: Resting BP; urine sample (female participants only); anthropometric measurements; high resolution ultrasound and carotid tonometry for measurement of arterial stiffness; pulse wave velocity; dispensing of placebo or fish oil supplement.

Visit 2: Resting BP; anthropometric measurements; high resolution ultrasound and carotid tonometry for measurement of arterial stiffness; pulse wave velocity; dispensing of placebo or fish oil supplement.

Visit 3: Resting BP; anthropometric measurements; high resolution ultrasound and carotid tonometry for measurement of arterial stiffness; pulse wave velocity; dispensing of placebo or fish oil supplement.

Visit 4: Resting BP; anthropometric measurements; high resolution ultrasound and carotid tonometry for measurement of arterial stiffness; pulse wave velocity; dispensing of placebo or fish oil supplement.

Note #1: If resting BP measurements are >130/80 mmHg during the first visit, the subject will be asked to schedule the session at least 48 hours later. If the resting BP measurements are >130/80 mmHg during the next visit, they will be excluded from the study and instructed to follow-up with their primary care provider.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-30 yearsa,d
2. Moderately active (exercise 3-5 days per week, >30 min per day)
3. Weight stable for previous 6 months (>2.5 kg)
4. Willing to be randomized to treatments and commit to all aspect of study
5. Provide health history questionnaire and informed consent.
6. Female subjects only- reported regular menstrual cycles for the last 2 years

Exclusion Criteria:

1. BP>140/90
2. Diabetes
3. Familial hypercholesterolemia
4. Past or current history of CHD, stroke or major CVD events. Respiratory diseases, endocrine or metabolic, neurological, or hematological disorders that would compromise the study or the health of the subject.
5. Active renal or liver disease
6. All medications that influence dependent variablesb
7. Recent surgery
8. Alcohol abusec
9. Women must not be pregnant, plan to become pregnant during the study, or be nursing
10. Claustrophobia

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Primary Aim | 6 weeks
  The primary outcome of the proposed study will be beta-stiffness which is calculated from maximal and minimal carotid diameters and carotid systolic and diastolic pressures.
Primary Aim | 6 weeks
  The secondary outcome of the proposed study will be pulse wave velocity which is measure of the time delay between the arrival of the pulse wave at the carotid and femoral arteries.

CONTACTS AND LOCATIONS:
Locations (1):
- Salisbury University, Salisbury, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided